CLINICAL TRIAL: NCT00345124
Title: The Effect of High and Low Sodium Intake on Urinary Aquaporin-2 in Essential Hypertension, During Basal Conditions and After Hypertonic Saline Infusion.
Brief Title: The Effect of High and Low Sodium Intake on Urinary Aquaporin-2 in Essential Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Carolina Cannillo Graffe, Department of Medical Research, Holstebro Hospital
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: med.res.hos.2006.cc.02
Record Dates: First submitted 2006-06-24; First posted 2006-06-27 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Essential Hypertension and Healthy Controls
Keywords: urinary aquaporin-2; ENaC; fractional sodium excretion; High/low sodium diet
MeSH Terms: conditions — Essential Hypertension | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: high sodium diet — 250-350 mmol
  Other Names: For four days
Behavioral: Low Sodium Diet — 25-35 mmol
  Other Names: For four days

SUMMARY:
The aim of the study is to test the following hypotheses:

* that the function and/or regulation of AQP2 and/or ENaC in the principal cells is abnormal in essential hypertension.
* if an abnormal function of the principal cells is present in essential hypertension, this will become more pronounced at high and low sodium intake.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men and women
* Age 18-65 years
* Arterial hypertension
* Body mass index between 18.5 and 30 kg/m2

Exclusion Criteria:

* Secondary hypertension
* Isolated systolic hypertension
* History or clinical signs of AMI, atrial fibrillation, disease of the heart valves, or chronic heart failure.
* Malignant disease
* Prior apoplexy
* alcohol or drug abuse
* Drug use except antihypertensives and oral contraceptives
* Abnormal biochemical screening of the blood regarding: red and white blood count, s-creatinine (> 200 micromol/L), b-hemoglobin, p-Sodium, p- potassium, p-albumine, p-bilirubin, p-alanine aminotransferase, p-alkaline phosphatase, p-cholesterol and b-glucose.
* Abnormal screening of the urine regarding: Blood, albumine and glucose.
* abnormal electrocardiogram
* Blood donation within one month of the first examination day
* Unwillingness to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-05; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
u-AQP-2 | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
fractional sodium excretion | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
p-vasopressin | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
p-aldosterone | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.

SECONDARY OUTCOMES:
u-p-AQP-2 | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
u-ENaC(alfa,beta,gamma) | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
CH2O | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
u-cAMP | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
uPGE2 | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
GFR | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Erling B. Pedersen, Professor, Study Chair — Department of Medical Research, Holstebro Hospital, Denmark; Carolina C. Graffe, MD, Principal Investigator — Department of Medical Research, Holstebro Hospital, Denmark
Locations (1):
- Department of Medical Research, Holstebro Hospital, Holstebro, Denmark

REFERENCES:
- [Derived] Graffe CC, Bech JN, Lauridsen TG, Vase H, Pedersen EB. Abnormal increase in urinary aquaporin-2 excretion in response to hypertonic saline in essential hypertension. BMC Nephrol. 2012 Mar 27;13:15. doi: 10.1186/1471-2369-13-15. PMID 22452789